CLINICAL TRIAL: NCT01195090
Title: Efficacy of Adding Sitagliptin or Pioglitazone to Patients With Type 2 Diabetes Insufficiently Controlled With Metformin and Sulfonylurea
Brief Title: Adding Sitagliptin or Pioglitazone to Type 2 Diabetes Mellitus Insufficiently Controlled With Metformin and Sulfonylurea
Acronym: JAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sung-Chen Liu (Other)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Sung-Chen Liu, Mackay Memorial Hospital, Mackay Memorial Hospital
Organization: Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09MMHIS047
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes
Keywords: sitagliptin; pioglitazone; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sitagliptin (Active Comparator): add sitagliptin100mg/d to pre-study OADs
  Interventions: Drug: Sitagliptin
- pioglitazone (Active Comparator): add pioglitazone 30mg/d to pre-study OADs
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: Sitagliptin — add sitagliptin100mg/d to pre-study OADs
  Other Names: Januvia
  Arms: sitagliptin
Drug: pioglitazone — add pioglitazone 30mg/d to pre-study OADs
  Other Names: actos
  Arms: pioglitazone

SUMMARY:
This 24-weeks study will to compare the glycemic efficacy and safety of sitagliptin with pioglitazone in patients with type 2 diabetes who had inadequate glycemic control despite dual therapy with metformin and a sulfonylurea.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, parallel, 24-week study. Inclusion criteria: type 2 diabetes patients who were treated with stable doses of sulfonylurea and metformin to their half maximally dose (sulfonylureas > half maximal dose, and metformin > 1500 mg/d) for > 10 weeks. > 20 years old; A1C:> 7.0 % and < 11% Exclusion criteria: insulin use within 12 weeks of the screening visit, any contraindications for use of sitagliptin or pioglitazone, impaired renal function (serum creatinine > 1.4 mg/dl), alanine aminotransferase (ALT) or aspartate aminotransferase levels (AST) > 2.5 times the upper limit of normal (ULN), current or prepare to pregnancy and lactation.

Primary Purpose:

compare the change in hemoglobin A1c and the proportion of patients achieving A1C < 7% between the 2 groups

Secondary Purposes:

1. Changes in fasting plasma glucose, high sensitive C-reactive protein (hsCRP)
2. Homeostasis model assessment-β cell function(HOMA-β) will be calculated to assess changes in β-cell function and HOMA-insulin resistance(HOMA-IR)to assess changes in insulin resistance
3. Body weight change, proportion of side effects

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients who were treated with stable doses of sulfonylurea and metformin to their half maximally dose (sulfonylureas > half maximal dose, and metformin > 1500 mg/d) for > 10 weeks
* > 20 years old
* A1C: > 7.0 % and < 11%

Exclusion Criteria:

* Insulin use within 12 weeks of the screening visit
* Any contraindications for use of sitagliptin or pioglitazone, impaired renal function (serum creatinine > 1.4 mg/dl), alanine aminotransferase or aspartate aminotransferase levels > 2.5 times the upper limit of normal
* Current or prepare to pregnancy and lactation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chen Liu, MD, Principal Investigator — Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was started from 01 OCT 2009 to 27 SEP 2011
Pre-assignment Details: we screened 135 patients and 120 patients were randomized in a 1: 1 ratio to one of the treatment groups.
  reson for excluded: 4 patients: ALT or AST >2.5x ULN 8 patiens : withdraw informed consent 3 patiens: baseline A1C>11%
Period: Overall Study
Arm/Group | Sitagliptin | Pioglitazone
Started | 60 | 60
Completed | 54 | 52
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Pioglitazone | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 49 | 91
  >=65 years | 18 | 11 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (8.9) | 58.1 (8.3) | 59.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 22 | 23 | 45
Region of Enrollment [Number; unit: participants]
  Taiwan | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Glycosylated Hemoglobin (A1C)
Description: A1C change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy.
Measure: Least Squares Mean (Standard Error); unit: percentage of Hb
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage of Hb | -0.71 (0.12) | -0.94 (0.12)
Statistical Analysis 1: Comparison: Sitagliptin vs Pioglitazone; The change from baseline in A1C were determined using an analysis of co-variance (ANCOVA) model with the factor 'treatment' and baseline A1C as covariate; Test type: Superiority or Other; p = 0.165, ANCOVA — The change from baseline in A1C were determined using an analysis of co-variance (ANCOVA) model with the factor 'treatment' and baseline A1C as covariate; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.58 to 0.08], Standard Error of Mean 0.16

2. Secondary Outcome: Changes in Fasting Plasma Glucose
Description: fasting serum sugar change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat (ITT) analysis with last observation carried forward was used to assess efficacy.
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | -23 (4.0) | -36 (4.0)

3. Secondary Outcome: Changes in High Sensitive C-reactive Protein
Description: fasting high sensitive serum C-reactive protein change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | -0.07 (0.04) | -0.19 (0.04)

4. Secondary Outcome: Changes in Homoeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy
Measure: Least Squares Mean (Standard Error); unit: HOMA-IR score
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
HOMA-IR score | -0.00 (0.35) | -1.56 (0.35)

5. Secondary Outcome: Body Weight Change
Description: body weight change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
kg | -0.26 (0.32) | 1.34 (0.32)

6. Secondary Outcome: Percentages of Patients With Total Adverse Events (AE)
Description: percentages of total adverse events
Time Frame: 24 weeks
Population: All patients who had taken at least one dose of study medication were included in the safety analysis
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 43.1 | 51.7

7. Secondary Outcome: Change in Fasting Total-cholesterol
Description: Total-cholesterol change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy.
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | 0.6 (3.9) | 9.9 (4.0)

8. Secondary Outcome: Change in Fasting Low-density Lipoprotein Cholesterol (LDL-C)
Description: LDL-C change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | -1.2 (3.7) | 6.6 (3.7)

9. Secondary Outcome: Change in Fasting Triglycerides(TG)
Description: TG change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy.
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | 6.3 (9.3) | -23.9 (9.4)

10. Secondary Outcome: Change in Fasting High-density Lipoprotein Cholesterol(HDL-C)
Description: HDL-C change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy.
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
mg/dl | 1.3 (1.2) | 6.3 (1.2)

11. Secondary Outcome: Change in Fasting Plasma Alanine-aminotransferase (ALT)
Description: ALT change from baseline to 24 weeks
Time Frame: 24 weeks
Population: An intent-to-treat analysis with last observation carried forward was used to assess efficacy
Measure: Least Squares Mean (Standard Error); unit: IU/L
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
IU/L | -0.0 (2.4) | -4.5 (2.4)

12. Secondary Outcome: Percentages of Patients With Mild to Moderate Hypoglycemia
Description: Incidence of mild to moderate hypoglycemia after treatment
Time Frame: 24 weeks
Population: All patients who had taken at least one dose of study medication were included in the safety analysis
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 10 | 8.5

13. Secondary Outcome: Percentages of Patients With Edema
Description: proportion of edema after treatment
Time Frame: 24 weeks
Population: All patients who had taken at least one dose of study medication were included in the safety analysis
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 0 | 27.1

14. Secondary Outcome: Percentages of Patients With Gastrointestinal Adverse Events
Description: Proportion of Gastrointestinal adverse events after treatment
Time Frame: 24 weeks
Population: All patients who had taken at least one dose of study medication were included in the safety analysis
Measure: Number; unit: percentge
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentge | 20.0 | 6.8

15. Secondary Outcome: Percentages of Patients With Nasopharyngitis
Description: Proportion of Nasopharyngitis after treatment
Time Frame: 24 weeks
Population: All patients who had taken at least one dose of study medication were included in the safety analysis
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 20.0 | 18.6

16. Primary Outcome: Baseline A1C
Description: baseline A1C
Time Frame: Baseline
Population: baseline Laboratory measurements
Measure: Mean (Standard Deviation); unit: percentage of Hb
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
percentage of Hb | 8.27 (0.86) | 8.54 (0.97)

17. Primary Outcome: The Percentages of Patient Achieving an A1C <7%
Description: The percentages of patient achieving an A1C <7% at endpoint
Time Frame: 24 weeks
Population: The percentages of patient achieving an A1C <7% at endpoint
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 28.3 | 28.8
Statistical Analysis 1: Comparison: Sitagliptin vs Pioglitazone; Chi-square test for percentages of patient achieving an A1C <7%; Test type: Non-Inferiority or Equivalence — Chi-square test; p = 0.954, Chi-squared — Chi-square test; Chi-Square = 0.0034

18. Secondary Outcome: Percentages of Patients With Severe Hypoglycemia
Description: Proportion of severe hypoglycemia after treatment
Time Frame: 24 weeks
Population: Proportion of severe ypoglycemia after treatment
Measure: Number; unit: percentage
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 59
percentage | 0 | 0

19. Secondary Outcome: Baseline Fasting Plasma Glucose
Description: Baseline fasting plasma glucose
Time Frame: baseline
Population: Baseline fasting plasma glucose
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 177 (47) | 182 (38)

20. Secondary Outcome: Baseline High Sensitive C-reactive Protein
Description: Baseline high sensitive C-reactive Protein
Time Frame: baseline
Population: Baseline high sensitive C-reactive Protein
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 0.38 (0.36) | 0.42 (0.68)

21. Secondary Outcome: Baseline Homoeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Baseline HOMA-IR
Time Frame: Baseline HOMA-IR
Population: Baseline HOMA-IR
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
HOMA-IR score | 5.6 (3.8) | 4.8 (3.2)

22. Secondary Outcome: Baseline Alanine-aminotransferase (ALT)
Description: Baseline alanine-aminotransferase
Time Frame: Baseline
Population: Baseline alanine-aminotransferase
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
IU/L | 34.2 (17.5) | 28.5 (15.5)

23. Secondary Outcome: Baseline Body Weight
Description: Baseline body weight
Time Frame: Baseline
Population: Baseline body weight
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
kg | 69.4 (13.6) | 65.4 (10.4)

24. Secondary Outcome: Baseline Total Cholesterol
Description: Baseline Total cholesterol
Time Frame: Baseline
Population: Baseline Total cholesterol
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 174 (31) | 194 (33)

25. Secondary Outcome: Baseline Triglyceride (TG)
Description: Baseline TG
Time Frame: Baseline
Population: Baseline TG
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 137 (74) | 164 (73)

26. Secondary Outcome: Baseline Low-density Lipoprotein Cholesterol (LDL-C)
Description: Baseline LDL-C
Time Frame: Baseline
Population: Baseline LDL-C
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 102 (25) | 111 (31)

27. Secondary Outcome: Baseline High-density Lipoprotein Cholesterol (HDL-C)
Description: Baseline HDL-C
Time Frame: Baseline
Population: Baseline HDL-C
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin | Pioglitazone
Number analyzed (Participants) | 60 | 60
mg/dl | 42 (12) | 43 (12)

ADVERSE EVENTS:
Time Frame: adverse event was recorded after 12 weeks and 24 weeks treatment or was recorded if adverse event was noted at any time during the study period.
Description: All adverse events was recorded after treatment. Symptomatic hypoglycemia was defined as an event with clinical symptoms consistent with hypoglycemia and severe hypoglycemia was defined as an event with symptoms consistent with hypoglycemia in which the patient required the assistance of another person.
Arm/Group | Sitagliptin | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 26/60 | 31/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=60) | Pioglitazone (N=60)
edema (General disorders) | 0 (0) | 16 (16) — 12 patients in the pioglitazone group had peripheral edema after treamtnet for 12 weeks and 16 patients had edema after treatment for 24 weeks. No edema in the sitagliptin group was noted.
Hypoglycemia (General disorders) | 6 (6) | 5 (5) — Hypoglycemic events occurred in 5 patients in the pioglitazone group and in 6 patients in the sitagliptin group. All the adverse events were mild to moderate.
Gastrointestinal adverse event (Gastrointestinal disorders) | 12 (12) | 4 (4) — Gastrointestinal adverse event was recorded at any visit after treatment
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 11 (11) — Nasopharyngitis was recorded at every visit

LIMITATIONS AND CAVEATS:
The reasons for withdrawal:

lost to follow-up:2 in pioglitazone and 2 in sitagliptin protocol violation:4 in pioglitazone and 3 in sitagliptin edema:1 in pioglitazone, ALT >3 times ULN:1 in pioglitazone gastrointestinal events:1 in sitagliptin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No